CLINICAL TRIAL: NCT05644821
Title: Influence of Electronic Patient Reported Outcomes (ePROMs) in Surgical Therapy for Prostate Cancer on Postoperative Outcome
Acronym: PRO-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Marienhospital Herne (Other); University Hospital, Essen (Other); University Hospital, Bonn (Other); Klinikum Dortmund gGbmH (Unknown); University Hospital Muenster (Other); University Hospital of Cologne (Other); University of Cologne (Other); Techniker Krankenkasse (Other); Deutsche Krebsgesellschaft e.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-2148
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Intention-to-treat principle, comparison (regarding superiority) of primary endpoint using mixed linear model for repeated measures: dependent variable: primary endpoint, influencing factors: Indicator for intervention/control group, time, group*time, center, tumor stage, and age group; downstream sequential-rejection testing of equality of expected values in the individual strata via appropriate contrasts; control of multiple error for at least one false rejection (final test principle); supplementary: mixed linear models with additional independent variables; sensitivity analyses on the influence of missing values (multiple imputation); subgroup analyses according to center, stage, and age group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group (Experimental): Patients who are not fully continent 6-weeks post-surgery (i.e., do not use pads in 24 hours) are randomized into the intervention or control group. In the intervention group, when the respective questionnaire thresholds are exceeded in the ePROM survey, an alarm is triggered at the treating prostate cancer center and contact is made by the center, as well as subsequent actions, if necessary.
  Interventions: Other: complex intervention
- Control group (No Intervention): Patients who are not fully continent 6-weeks post-surgery (i.e., do not use pads in 24 hours) are randomized into the intervention or control group. In the control group, ePROMs will be collected 24 and 52 weeks after radical prostatectomy, but without triggering an alarm with subsequent measures - the control group will therefore receive treatment according to the current clinical routine.
- Comparison group (Other): In patients who are fully continent 6-weeks post-surgery (i.e., do not use pads in 24 hours), ePROMs are collected at 24 and 52 weeks, but no alarms or further actions are derived from them. Thus, treatment is provided according to routine clinical practice. Patients are not randomized.
  Interventions: Other: current clinical practice

INTERVENTIONS:
Other: complex intervention — The intervention has several elements:
  1. Regular symptom monitoring via ePROMs
  2. Alarm when defined thresholds of EPIC-26 or PHQ-4 are reached or exceeded, 3.) In case of alarm, standardized telephone contact by a study nurse at the treating center with the offer to coordinate a urological consultation at the center, 4.) if requested by the patient: a urological consultation at the treating prostate cancer center by urologists trained in the PRO-P study,
  4) content of the consultation: if necessary, the guideline-compliant initiation of further diagnostics and therapy including in this context necessary follow-up contacts and 5) postal communication of the ePROM results in case of an alarm as well as postal dispatch of a report of the findings in case of a urological consultation at the treating prostate cancer center to the practicing, treating urologist.
  Arms: Intervention group
Other: current clinical practice — current clinical practice
  Arms: Comparison group

SUMMARY:
The study investigates the influence of structured follow-up using ePROMS in the 1st year after prostatectomy on the postoperative course. It will be examined whether this intervention leads to early detection of postoperative symptoms and whether the subsequent initiation of further measures lead to an improvement of incontinence, symptom burden, quality of life and patient competence.

DETAILED DESCRIPTION:
PRO-P is planned as a multicenter, prospective, and two-arm randomized control group study in which ePROMs will be performed in a standardized fashion once before and six times (intervention group) or three times (control group) after primary prostatectomy in patients with PCa. PROMs are collected either web-based or through a dedicated app and entered by the patient using either a mobile device or computer. Patients are invited to enter ePROMS into the app or web tool through email and app-driven push messages. Patients who are incontinent (at least one pad in 24 hours) at the 6-week postoperative survey are randomized into two groups: The intervention group and the control group. In the intervention group, when the respective questionnaire cut-off values are exceeded in the ePROM survey, an alarm is triggered at the treating prostate cancer center and contact is made by the center as well as subsequent measures, if necessary. This is done at 6 weeks postoperatively and at 12, 18, 24, 36 and 52 weeks postoperatively. In the control group, ePROMs are recorded 24 and 52 weeks after radical prostatectomy, but without triggering an alarm with subsequent measures - the control group thus receives treatment in accordance with the current clinical routine. The mechanisms of action of the intervention will be investigated within the framework of a qualitative process evaluation. Characteristics on the patient level (e.g., treatment-related attitudes, comorbidity, social support), on the practitioner level (e.g., communication skills), on the organizational level, and the interactions between the levels (e.g., patient-doctor relationship) will be explored. The goal is to develop an intervention model, or to describe the effective elements of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 y
* legal capacity
* sufficient knowledge of the German language
* prostate carcinoma, TNM T1-4 NX N0-1 M0-1c
* primary radical prostatectomy planned
* mobile input device or PC available
* ability to either receive emails or install a special app on cell phone and receive push messages, with guidance or assistance if necessary
* ability to complete electronic questionnaires, with guidance or assistance if necessary

Exclusion Criteria:

* palliative treatment situation (life expectancy < 1 year)
* preoperative urinary incontinence (at least one pad per 24 hours)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
urinary incontinence | 52 weeks
  The Expanded Prostate Cancer Index Short Form (EPIC-26) is a questionnaire that assesses symptoms and functions of people with prostate cancer in 5 domains. A total of 100 points can be achieved for each domain, with a higher score indicating better function. The urinary incontinence domain consists of four items. To calculate the primary endpoint, the difference between the scores on the urinary incontinence scale of the EPIC-26 is taken at 52 and 6 weeks. Changes regarding urinary incontinence (Minimally Important Difference (MID) >= 9) at 52 weeks postoperatively compared with 6 weeks postoperatively are considered.

SECONDARY OUTCOMES:
EPIC-26: changes in sexual function | 52 weeks
  Similar to the primary endpoint, changes at 52 weeks postoperatively compared with 6 weeks postoperatively are considered for the changes in in sexual function according to EPIC-26 (MID >= 10).
EPIC-26: changes in irritative/obstructive symptoms | 52 weeks
  Similar to the primary endpoint, changes at 52 weeks postoperatively compared with 6 weeks postoperatively are considered for the changes in irritative/obstructive an gastrointestinal symptoms according to EPIC-26 (MID >= 7).
EPIC-26: changes in gastrointestinal symptoms | 36 months
  Similar to the primary endpoint, changes at 52 weeks postoperatively compared with 6 weeks postoperatively are considered for the changes an gastrointestinal symptoms according to EPIC-26 (MID >= 5).
EPIC-26: changes in vitality/hormonal function | 52 weeks
  Similar to the primary endpoint, changes at 52 weeks postoperatively compared with 6 weeks postoperatively are considered for the changes in vitality/ hormonal function according to EPIC-26 (MID >= 4).
EQ-5D-5L: changes in health-related quality of life (HRQoL) | 52 weeks
  The European Quality of Life Five-Dimensions Questionnaire (EQ-5D-5L) measures health-related quality of life on five scales: 1. mobility, 2. ability to care for oneself, 3. activities of daily living, 4. pain/physical discomfort, and 5. anxiety/dejection, each of which is represented by a question that provides five response options for grading symptoms. In addition, a question on self-assessment of health status is asked on a visual analog scale from 0 to 100, where 100 is the best imaginable health.
PHQ-4: changes in depressivity | 52 weeks
  The Patient Health Questionnaire-4 (PHQ-4) measures depressiveness and generalized anxiety on two subscales with two items each. For each question, scores from 0 to 3 can be achieved, so that a cumulative score of 12 points can be reached, whereby a higher score indicates a more pronounced symptomatology. The cut-off value for depressivity is defined for the subscales of the PHQ-4 is definied by >= 3 points, the respective attainment of which (independent of the preoperative value) triggers an alarm at each survey time point.
PHQ-4: changes in generalised anxiety | 52 weeks
  The Patient Health Questionnaire-4 (PHQ-4) measures depressiveness and generalized anxiety on two subscales with two items each. For each question, scores from 0 to 3 can be achieved, so that a cumulative score of 12 points can be reached, whereby a higher score indicates a more pronounced symptomatology. The cut-off value for depressivity is defined for the subscales of the PHQ-4 is definied by >= 3 points, the respective attainment of which (independent of the preoperative value) triggers an alarm at each survey time point.
PEI: changes in patient enablement | 52 weeks
  The Patient Enablement Instrument (PEI) measures patient empowerment through six questions; a validated German translation with a modified question sequence and Likert scale is used. Overall, the sum score ranges from 6 to 30 points, with a higher score corresponding to greater patient empowerment.
qualitative process evaluation - module 1: feasibility | 52 weeks
  semi-structured interviews with patients, urologists, psychooncologists, study nurses (N=10-15); data from Module 1 will be evaluated qualitatively using content analysis; criteria are based on the feasibility criteria for evaluating the acceptance and feasibility of the intervention and the study procedures
qualitative process evaluation - module 2: impact | 52 weeks
  sequential semi-structured interviews with patients and relatives from the intervention and control groups in the main study (N=30-40); data from module 2 will be evaluated by contrastive thematic coding; in addition to possible differences between the intervention and control groups, intraindividual changes are also evaluated by contrastive coding of the data material at several time points
qualitative process evaluation - module 3: implementation | 52 weeks
  Semi-structured interviews with urologists, psychooncologists, study nurses in the main study (N=10-15); focus group discussion with study participants; analysis of implementation factors is guided by the Consolidated Framework for Advancing Implementation Science (CFIR); data from module 3 on implementation are evaluated qualitatively by content analysis

CONTACTS AND LOCATIONS:
Overall Officials: Peter Albers, MD, Principal Investigator — University Clinic Düsseldorf, Urology; André Karger, MD, Study Director — University Clinic Düsseldorf, psychosomatic medicine
Locations (5):
- Germany (5):
  - University Clinic Bonn, Urology, Bonn, North Rhine Westpahlia
  - Klinikum Dortmund gGmbH, Urology, Dortmund, North Rhine-Westphalia
  - University Clinic Düsseldorf, Urology, Düsseldorf, North Rhine-Westphalia
  - University Clinik Bochum, Marienhospital Herne, Urology, Herne, North Rhine-Westphalia
  - University Clinic Münster, Urology, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Monajjed R, Albers P, Droop J, Fugmann D, Noldus J, Palisaar RJ, Ritter M, Ellinger J, Krausewitz P, Truss M, Hadaschik B, Grunwald V, Schrader AJ, Papavassilis P, Ernstmann N, Schellenberger B, Moritz A, Kowalski C, Hellmich M, Heiden P, Hagemeier A, Horenkamp-Sonntag D, Giessing M, Pauler L, Dieng S, Peters M, Feick G, Karger A; PRO-P study group. PRO-P: evaluating the effect of electronic patient-reported outcome measures monitoring compared with standard care in prostate cancer patients undergoing surgery-study protocol for a randomized controlled trial. Trials. 2024 Nov 12;25(1):754. doi: 10.1186/s13063-024-08579-8. PMID 39533412